CLINICAL TRIAL: NCT01615952
Title: Patient Positioning on Supraclavicular Nerve Block
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Antoun Nader, Professor of Anesthesiology, Northwestern University
Other Study IDs: STU00058413; Northwestern University
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Nerve Block
Keywords: Supraclavicular Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Sitting Position (head of bed 90 degrees): Ultrasound measurements will be performed. A= skin to the pleura at the level lateral to the subclavian artery, B= skin to center of the subclavian artery, C= skin to first rib, D= skin to "corner pocket"
- Semi-sitting position (45 degrees): Ultrasound measurements will be performed. A= skin to the pleura at the level lateral to the subclavian artery, B= skin to center of the subclavian artery, C= skin to first rib, D= skin to "corner pocket"
- Supine position: Ultrasound measurements will be performed. A= skin to the pleura at the level lateral to the subclavian artery, B= skin to center of the subclavian artery, C= skin to first rib, D= skin to "corner pocket"

SUMMARY:
Blockade of the brachial plexus using a supraclavicular approach provides excellent anesthesia for upper extremity surgery. The most serious complication specific to this block is pneumothorax. Subsequent modifications of this block including the use of ultrasound have lowered the risk from 6% to <1%. Case reports remain and authors have described certain factors and strategies to reduce this risk. Most texts and journals describe the patient in a supine or semi-sitting position during the block. At the investigators institution the investigators perform the block in a semi-sitting position to facilitate needle tip visibility with ultrasound. The investigators plan to obtain ultrasound anatomic measurements in three different positions (supine, semi-sitting, sitting) using patients consented for supraclavicular nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* all patients, 18 y/o to 65 y/o, who are scheduled to receive an ultrasound- guided supraclavicular nerve block

Exclusion Criteria:

* patient refusal to be included in the study,
* the presence of language barrier that inhibits proper communication with the patient, contraindications to regional anesthesia (local infection, severe pulmonary disease, or preexisting neuropathy)
* history of allergy to amide local anesthetics or narcotics
* the presence of a progressive neurological deficit
* history of hepatorenal insufficiency
* the presence of a coagulopathy or infection
* pregnancy
* a history of psychiatric disorder
* inability to follow study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 y/o to 65 y/o, who are scheduled to receive a ultrasound-guided supraclavicular nerve block as part of their postoperative pain management.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
patient positioning | Postoperative Day One
  Ultrasound measurements will be made at three different positions: Sitting, semi-sitting, and supine. The ultrasound measurements include A= skin to the pleura at the level lateral to the subclavian artery, B= skin to center of the subclavian artery, C= skin to first rib, D= skin to "corner pocket"

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feingberg School of Medicine, Chicago, Illinois, United States